CLINICAL TRIAL: NCT03371719
Title: A Phase II, Double-Blinded, Placebo-Controlled Randomized Trial of Salvage Radiotherapy With or Without Enhanced Anti-Androgen Therapy With Apalutamide in Recurrent Prostate Cancer (BALANCE*)
Brief Title: Radiation Therapy With or Without Apalutamide in Treating Patients With Recurrent Prostate Cancer, the BALANCE Trial
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NRG Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NRG-GU006; NCI-2017-01268 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-GU006 (Other: NRG Oncology); NRG-GU006 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2017-12-08; First posted 2017-12-13 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Recurrent Prostate Carcinoma; Stage III Prostate Adenocarcinoma AJCC v7; Stage IV Prostate Adenocarcinoma AJCC v7
MeSH Terms: conditions — Prostatic Neoplasms | interventions — apalutamide; Congresses as Topic; Radiation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (radiation therapy, placebo) (Active Comparator): Patients undergo external beam radiation therapy on day 1 for 7-8 weeks. Beginning on day of radiation therapy, patients receive placebo PO QD on days 1-30. Treatment repeats every 30 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: External Beam Radiation Therapy; Other: Placebo Administration
- Arm 2 (radiation therapy, apalutamide) (Experimental): Patients undergo external beam radiation therapy on day 1 for 7-8 weeks. Beginning on day of radiation therapy, patients receive apalutamide PO QD on days 1-30. Treatment repeats every 30 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Apalutamide; Radiation: External Beam Radiation Therapy

INTERVENTIONS:
Drug: Apalutamide — Given PO
  Other Names: ARN 509; ARN-509; ARN509; Erleada; JNJ 56021927; JNJ-56021927
  Arms: Arm 2 (radiation therapy, apalutamide)
Radiation: External Beam Radiation Therapy — Undergo external beam radiation therapy
  Other Names: Definitive Radiation Therapy; EBRT; External Beam Radiation; External Beam Radiotherapy; External Beam Radiotherapy (conventional); External Beam RT; external radiation; External Radiation Therapy; external-beam radiation; Radiation, External Beam; Teleradiotherapy; Teletherapy; Teletherapy Radiation
Other: Placebo Administration — Given PO
  Arms: Arm 1 (radiation therapy, placebo)

SUMMARY:
This phase II trial studies how well radiation therapy with or without apalutamide works in treating patients with prostate cancer that has come back (recurrent). Radiation therapy uses high energy x-ray to kill tumor cells and shrink tumors. Androgen can cause the growth of prostate cancer cells. Drugs, such as apalutamide, may lessen the amount of androgen made by the body. Giving radiation therapy and apalutamide may work better at treating prostate cancer compared to radiation therapy alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine whether, in men with post-prostatectomy prostate-specific antigen (PSA) recurrences, salvage radiation (SRT) with enhanced anti-androgen therapy with apalutamide will improve biochemical progression-free survival (bPFS) compared to SRT alone.

SECONDARY OBJECTIVES:

I. To assess whether molecular stratification by the PAM50 gene expression clustering will identify subsets of prostate cancer (luminal A or basal, luminal B) which derive the greatest benefit from anti-androgen therapy.

II. To assess overall survival. III. To assess cancer-specific mortality. IV. To assess metastasis-free survival. V. To assess distant metastasis. VI. To assess local-regional progression. VII. To assess PSA nadir during first year of treatment and prior to initiation of any hormonal salvage therapy.

VIII. To assess initiation of salvage hormonal therapy. IX. To assess PSA with a non-castrate testosterone at 1 and 3 years post randomization: PSA < 0.1 ng/ml and testosterone >= 50 ng/dl.

X. To assess acute and late physician-reported morbidity (per the Common Terminology Criteria for Adverse Events [CTCAE] version 5.0) after SRT +/- apalutamide.

XI. To assess acute and late patient-reported symptomatic adverse events morbidity (per the patient reported outcomes [PRO]-CTCAE) after SRT +/- apalutamide.

XII. To assess testosterone levels at 3, 6, 9, 12, and 36 months post randomization.

EXPLORATORY OBJECTIVE:

I. To assess the prognostic and predictive value of the genomic classifier Decipher.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM 1: Patients undergo external beam radiation therapy on day 1 for 7-8 weeks. Beginning on day of radiation therapy, patients receive placebo orally (PO) once daily (QD) on days 1-30. Treatment repeats every 30 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.

ARM 2: Patients undergo external beam radiation therapy on day 1 for 7-8 weeks. Beginning on day of radiation therapy, patients receive apalutamide PO QD on days 1-30. Treatment repeats every 30 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years, then every 6 months for 3 years, and then yearly thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histologically) proven diagnosis of prostate adenocarcinoma; prostatectomy must have been performed within 10 years prior to Step 1 registration and any type of radical prostatectomy is permitted, including retropubic, perineal, laparoscopic or robotically assisted
* Post-prostatectomy patients with a detectable serum PSA (>= 0.1, but =< 1.0 ng/mL) at study entry (within 90 days of Step 1 registration) and at least one of the following:

  * Gleason score 7-10 (International Society of Urological Pathology [ISUP] grade group 2 to 5)
  * ISUP grade group:

    * Grade group 1 = Gleason score =< 6,
    * Grade group 2 = Gleason score 3 + 4 = 7,
    * Grade group 3 = Gleason score 4 + 3 = 7,
    * Grade group 4 = Gleason score 8,
    * Grade group 5 = Gleason scores 9 and 10
  * >= T3a disease
  * Persistent elevation of PSA after prostatectomy measured within 90 days after surgery (PSA never became undetectable) of > 0.04 but < 0.2 ng/mL (PSA nadir)
* pN0 or pNx
* History/physical examination within 90 days prior to Step 1 registration
* Karnofsky performance status of 70-100 within 90 days prior to Step 1 registration
* Surgical formalin-fixed paraffin-embedded (FFPE) specimen must be available for submission to GenomeDx for genomic analysis on Decipher GRID platform; Note: if Decipher results have already been obtained, in lieu of tissue, results must be submitted to GenomeDx for validation and for GenomeDx to provide the subtyping needed for stratification
* Prior androgen deprivation therapy (luteinizing hormone-releasing hormone [LHRH] agonist and/or non-steroidal anti-androgen) is allowed if discontinued at least 90 days prior to Step 1 registration and given for =< 90 days duration

  * For example: patients on prior LHRH analogs (post-prostatectomy), the discontinuation date should be calculated based on the expected duration of the sustained release injection, not simply the injection date of the drug; for instance, if a 22.5 mg sustained release dose of leuprolide acetate is given (3 month duration), then the expected duration of such a dose would be 90 days after the injection date; for a 7.5 mg leuprolide (1 month duration), the discontinuation date would be 30 days after the injection date
  * Please note: finasteride or dutasteride must be stopped before treatment starts but prior usage will not affect eligibility
* Hemoglobin >= 9.0 g/dL, independent of transfusion and/or growth factors within 90 days prior to Step 1 registration
* Platelet count >= 100,000 x 10^9/uL independent of transfusion and/or growth factors within 90 days prior to Step 1 registration
* Serum albumin >= 3.0 g/dL within 90 days prior to Step 1 registration
* Glomerular filtration rate (GFR) >= 35 mL/min estimated by Cockcroft-Gault or measured directly by 24 hour urine creatinine within 90 days prior to Step 1 registration
* Serum total bilirubin =< 1.5 x upper limit of normal (ULN) (Note: in subjects with Gilbert's syndrome, if total bilirubin is > 1.5 x ULN, measure direct and indirect bilirubin and if direct bilirubin is =< 1.5 x ULN, subject is eligible) within 90 days prior to Step 1 registration
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) < 2.5 x ULN within 90 days prior to Step 1 registration
* Testosterone > 50 ng/dL within 90 days prior to Step 1 registration
* Concomitant medications known to lower the seizure threshold discontinued or substituted at least 4 weeks (30 days) prior to Step 1 registration
* The patient must agree to use a condom (even men with vasectomies) and another effective method of birth control if he is having sex with a woman of childbearing potential or agree to use a condom if he is having sex with a woman who is pregnant while on study drug and for 3 months following the last dose of study drug
* The patient must agree not to donate sperm during the study treatment and for 3 months after receiving the last dose of study drug
* The patient or a legally authorized representative must provide study-specific informed consent prior to study entry

Exclusion Criteria:

* PRIOR TO STEP 1 REGISTRATION:
* Definitive clinical, radiologic, or pathologic evidence of metastatic disease (M1) or lymph node involvement (N1)
* Prior invasive malignancy (except non-melanomatous skin cancer, carcinoma in situ of the male breast, penis, oral cavity, or stage Ta of the bladder, or stage I completely resected melanoma) unless disease free for a minimum of 2 years
* Prior systemic chemotherapy for the study cancer; note that prior chemotherapy for a different cancer is allowable
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields
* History of any of the following:

  * Seizure or known condition that may pre-dispose to seizure (e.g. prior stroke within 1 year prior to Step 1 registration)
  * History of documented inflammatory bowel disease
  * Transmural myocardial infarction within the last 4 months prior to Step 1 registration
  * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months prior to Step 1 registration
  * History of any condition that in the opinion of the investigator, would preclude participation in this study
* Current evidence of any of the following:

  * Known gastrointestinal disorder affecting absorption of oral medications
  * Active uncontrolled infection (e.g., human immunodeficiency virus [HIV] or viral hepatitis)
  * Uncontrolled hypertension
  * Any current condition that in the opinion of the investigator, would preclude participation in this study
* Prior whole gland ablative therapy (i.e. cryoablation or high intensity focused ultrasound [HIFU]) for prostate cancer is not allowed
* HIV positive with CD4 count < 200 cells/microliter within 30 days prior to registration
* HIV patients under treatment with highly active antiretroviral therapy (HAART) within 30 days prior to registration regardless of CD4 count; (Note: HIV testing is not required for eligibility for this protocol as it is self-reported; this exclusion criterion is necessary because the treatments involved in this protocol may be immunosuppressive and/or interact with HAART)
* Patients must not plan to participate in any other clinical trials while receiving treatment on this study or being followed post-protocol therapy
* PRIOR TO STEP 2 REGISTRATION:
* For patients who have not undergone prior Decipher analysis, submission of the specimen to GenomeDx should be as soon as possible after study registration (Step 1) as these results can take up 21 days after the specimen is received at GenomeDx; Step 2 registration must occur within 6 weeks (42 days) of Step 1 registration; if Decipher results have already been obtained, in lieu of tissue, results must be submitted to GenomeDx for validation

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Estimated)
Dates: Start 2018-06-20 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Biochemical progression-free survival (bPFS) | From randomization to the first occurrence of a rise in PSA, clinical or radiographic local, regional, or distant metastases, or death from any cause, assessed up to 5 years
  bPFS curves will be estimated by the Kaplan-Meier (1958) method and compared between the two treatment arms using a one-sided logrank test at the alpha = 0.12 significance level. In addition, a multivariable Cox regression model will be fit incorporating the three stratification factors used in the randomization (surgical margins, pre-salvage radiation [SRT] PSA, and molecular subtype) as covariates to estimate the adjusted hazard ratio (HR) between the two treatment groups. Additional regression models will be fit including other pretreatment characteristics as covariates. The goodness-of-fit of the proportional hazards assumption will be evaluating using graphical methods (Kay, 1977), residual plots, and the global test proposed by Grambsch and Therneau (1994). Missing covariates will be handled using multiple imputation as described in White and Royston (1982).

SECONDARY OUTCOMES:
Overall survival (OS) | From randomization until death from any cause, assessed up to 5 years
  OS will be estimated by the Kaplan-Meier method and compared between treatment arms via the logrank test. Cox regression will be used to obtain HRs for this outcome, both unadjusted and adjusted for covariates.
Cancer-specific mortality (CSM) | From the date of randomization to the date of death due to prostate cancer, assessed up to 5 years
  CSM will be estimated by the Kaplan-Meier method and compared between treatment arms via the logrank test. Cox regression will be used to obtain HRs for this outcome, both unadjusted and adjusted for covariates. A competing risks analysis will be performed treating death from prostate cancer as the event of interest and death from all other causes as a competing risk. Cumulative incidence curves will be generated (Gooley et al., 1999; Dignam et al., 2004) along with 95% confidence intervals and compared between the two treatment arms using Gray's method (Gray, 1988). In addition, multivariable analysis will be conducted using Fine and Gray's regression model (Fine and Gray, 1999) to derive covariate-adjusted (subdistribution) HRs and confidence intervals.
Metastasis-free survival (MFS) | From randomization until distant metastasis (clinical and/or radiographic appearance of disseminated disease) or death from any cause, assessed up to 5 years
  MFS will be estimated by the Kaplan-Meier method and compared between treatment arms via the logrank test. Cox regression will be used to obtain HRs for this outcome, both unadjusted and adjusted for covariates. A competing risks analysis will be performed treating death from prostate cancer as the event of interest and death from all other causes as a competing risk. Cumulative incidence curves will be generated (Gooley et al., 1999; Dignam et al., 2004) along with 95% confidence intervals and compared between the two treatment arms using Gray's method (Gray, 1988). In addition, multivariable analysis will be conducted using Fine and Gray's regression model (Fine and Gray, 1999) to derive covariate-adjusted (subdistribution) HRs and confidence intervals.
Distant metastasis | Up to 5 years
  Will also be analyzed under a competing risks framework, treating death without experiencing the event in question as a competing risk.
Local-regional progression | From randomization to local or regional recurrence ignoring biochemical failure and distant recurrence and censoring for death, assessed up to 5 years
  Will also be analyzed under a competing risks framework, treating death without experiencing the event in question as a competing risk.
PSA nadir during first year of treatment and prior to initiation of any hormonal salvage therapy | During first year of treatment
  Will be compared between the two groups using a two-sample t-test.
Initiation of salvage hormonal therapy | Up to 5 years
  Will also be analyzed under a competing risks framework, treating death without experiencing the event in question as a competing risk.
Undetectable PSA with a non-castrate testosterone (PSA < 0.1 ng/ml and testosterone >= 50 ng/dl) | 1 year
  Will be compared using chi square tests.
Undetectable PSA with a non-castrate testosterone (PSA < 0.1 ng/ml and testosterone >= 50 ng/dl)) | 3 years
  Will be compared using chi square tests.
Acute physician-reported morbidity (per the Common Terminology Criteria for Adverse Events [CTCAE] version 5) | Up to 30 days after radiation therapy
  Adverse events will be scored according to the National Cancer Institute (NCI)'s CTCAE version 5.0. For each type of adverse event, counts and frequencies will be provided for the worst grade experienced by the patient by treatment arm. The proportion of patients with grades >= 1 and >= 3 will be compared between groups using a chi-square test, or Fisher's exact test if cell frequencies are < 5, at the two-sided 0.05 significance level. Logistic regression, both univariate and multivariate, will be used to model the probability of grade 3+ acute adverse events as a function of treatment arm and covariates. Both unadjusted and adjusted odds ratios and the respective 95% confidence intervals will be computed.
Late physician-reported morbidity (per the CTCAE version 5) defined as grade 3+ adverse events occurring more than 30 days after the completion of radiation therapy | From the time protocol treatment started to the time of the first recorded late grade 3+ adverse event, assessed up to 5 years
  Adverse events will be scored according to the NCI's CTCAE version 5.0. For each type of adverse event, counts and frequencies will be provided for the worst grade experienced by the patient by treatment arm. The proportion of patients with grades >= 1 and >= 3 will be compared between groups using a chi-square test, or Fisher's exact test if cell frequencies are < 5, at the two-sided 0.05 significance level.
Testosterone levels | Every 3 months until 6 months post treatment
  Testosterone levels will be assessed.
Acute patient-reported morbidity symptomatic adverse events (per the patient reported outcomes [PRO]-CTCAE) | Up to 5 years
  Adverse events will also be assessed using PRO-CTCAE items. Assessments will be collected before and at the end of radiotherapy treatment and in follow-up. For each symptom and each domain (i.e., frequency, severity, and interference), counts and frequencies will be provided for the worst score experienced by the patient by treatment arm. The proportion of patients with scores >= 1 and >= 3 will be compared between groups using a chi-square test, or Fisher's exact test if cell frequencies are < 5.
Late patient-reported morbidity symptomatic adverse events (per the PRO-CTCAE) | Up to 5 years
  Adverse events will also be assessed using PRO-CTCAE items. Assessments will be collected before and at the end of radiotherapy treatment and in follow-up. For each symptom and each domain (i.e., frequency, severity, and interference), counts and frequencies will be provided for the worst score experienced by the patient by treatment arm. The proportion of patients with scores >= 1 and >= 3 will be compared between groups using a chi-square test, or Fisher's exact test if cell frequencies are < 5.

CONTACTS AND LOCATIONS:
Overall Officials: Felix Y Feng, Principal Investigator — NRG Oncology
Locations (360):
- United States (352):
  - Arizona Center for Cancer Care - Gilbert, Gilbert, Arizona
  - Arizona Center for Cancer Care-Peoria, Peoria, Arizona
  - Arizona Center for Cancer Care - Scottsdale, Scottsdale, Arizona
  - Arizona Center for Cancer Care-Surprise, Surprise, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Marin General Hospital, Greenbrae, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Cancer Care and Hematology-Fort Collins, Fort Collins, Colorado
  - Valley View Hospital Cancer Center, Glenwood Springs, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - Stamford Hospital/Bennett Cancer Center, Stamford, Connecticut
  - Helen F Graham Cancer Center, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - AdventHealth Altamonte, Altamonte Springs, Florida
  - Regional Cancer Center-Lee Memorial Health System, Fort Myers, Florida
  - AdventHealth Kissimmee, Kissimmee, Florida
  - AdventHealth Orlando, Orlando, Florida
  - AdventHealth East Orlando, Orlando, Florida
  - Cleveland Clinic-Weston, Weston, Florida
  - AdventHealth Winter Park, Winter Park, Florida
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Edward Hines Jr VA Hospital, Hines, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - Parkview Regional Medical Center, Fort Wayne, Indiana
  - Goshen Center for Cancer Care, Goshen, Indiana
  - Reid Health, Richmond, Indiana
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - East Jefferson General Hospital, Metairie, Louisiana
  - LSU Healthcare Network / Metairie Multi-Specialty Clinic, Metairie, Louisiana
  - MaineHealth Coastal Cancer Treatment Center, Bath, Maine
  - MaineHealth Waldo Hospital, Belfast, Maine
  - MaineHealth Maine Medical Center - Biddeford, Biddeford, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - MaineHealth Stephens Hospital, Norway, Maine
  - MaineHealth Maine Medical Center - Portland, Portland, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - MaineHealth Cancer Care and IV Therapy - Sanford, Sanford, Maine
  - MaineHealth Cancer Care Center of York County, Sanford, Maine
  - MaineHealth Maine Medical Center- Scarborough, Scarborough, Maine
  - MaineHealth Cancer Care and IV Therapy - South Portland, South Portland, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Saint Agnes Hospital, Baltimore, Maryland
  - Central Maryland Radiation Oncology in Howard County, Columbia, Maryland
  - UM Baltimore Washington Medical Center/Tate Cancer Center, Glen Burnie, Maryland
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Michigan Healthcare Professionals Clarkston, Clarkston, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - Michigan Healthcare Professionals Farmington, Farmington Hills, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Michigan Healthcare Professionals Troy, Troy, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Mayo Clinic Health System in Albert Lea, Albert Lea, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Mayo Clinic Health Systems-Mankato, Mankato, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Minneapolis VA Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Kansas City Veterans Affairs Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Oncology Las Vegas - Henderson, Henderson, Nevada
  - Desert West Surgery, Las Vegas, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Hope Cancer Care of Nevada, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Oncology Las Vegas - Tenaya, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Solinsky Center for Cancer Care, Manchester, New Hampshire
  - Virtua Memorial, Mount Holly, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Sidney Kimmel Cancer Center Washington Township, Sewell, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - New Mexico Oncology Hematology Consultants, Albuquerque, New Mexico
  - New York-Presbyterian/Brooklyn Methodist Hospital, Brooklyn, New York
  - Sands Cancer Center, Canandaigua, New York
  - Mary Imogene Bassett Hospital, Cooperstown, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Wilmot Cancer Institute Radiation Oncology at Greece, Rochester, New York
  - Highland Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - James J Peters VA Medical Center, The Bronx, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Novant Cancer Institute Radiation Oncology - Supply, Supply, North Carolina
  - Novant Health Cancer Institute Radiation Oncology - Wilmington, Wilmington, North Carolina
  - Novant Health New Hanover Regional Medical Center, Wilmington, North Carolina
  - Summa Health System - Akron Campus, Akron, Ohio
  - Cleveland Clinic Akron General, Akron, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Geauga Hospital, Chardon, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - First Dayton Cancer Care, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Cleveland Clinic Cancer Center Mansfield, Mansfield, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - UH Seidman Cancer Center at Southwest General Hospital, Middleburg Heights, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - University Hospitals Portage Medical Center, Ravenna, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - UH Seidman Cancer Center at Firelands Regional Medical Center, Sandusky, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - Dayton Physicians LLC - Troy, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Cancer Treatment Centers of America, Tulsa, Oklahoma
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - UPMC Altoona, Altoona, Pennsylvania
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Northeast Radiation Oncology Center, Dunmore, Pennsylvania
  - UPMC Cancer Center at UPMC Horizon, Farrell, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - UPMC Cancer Center - Monroeville, Monroeville, Pennsylvania
  - UPMC Hillman Cancer Center in Coraopolis, Moon Township, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Jefferson Torresdale Hospital, Philadelphia, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - UPMC Uniontown Hospital Radiation Oncology, Uniontown, Pennsylvania
  - UPMC Washington Hospital Radiation Oncology, Washington, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - The Radiation Oncology Center-Hilton Head/Bluffton, Hilton Head Island, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - The West Clinic - Wolf River, Germantown, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Audie L Murphy VA Hospital, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Farmington Health Center, Farmington, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Riverton Hospital, Riverton, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Saint George Regional Medical Center, St. George, Utah
  - Southwestern Vermont Medical Center, Bennington, Vermont
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Dartmouth Cancer Center - North, Saint Johnsbury, Vermont
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - Hunter Holmes McGuire Veterans Administration Medical Center, Richmond, Virginia
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Froedtert Menomonee Falls Hospital, Menomonee Falls, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Zablocki Veterans Administration Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Froedtert West Bend Hospital/Kraemer Cancer Center, West Bend, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
- Canada (8):
  - Arthur J E Child Comprehensive Cancer Centre, Calgary, Alberta
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - CIUSSSEMTL-Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - The Research Institute of the McGill University Health Centre (MUHC), Montreal, Quebec
  - CHU de Quebec-L'Hotel-Dieu de Quebec (HDQ), Québec, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke-Fleurimont, Sherbrooke, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan